CLINICAL TRIAL: NCT00374075
Title: In Vivo Study of Safety, Tolerability and Dosing Effect on SMN mRNA and Protein Levels of Valproic Acid in Patients With Spinal Muscular Atrophy
Brief Title: Study of Safety and Dosing Effect on SMN Levels of Valproic Acid (VPA) in Patients With Spinal Muscular Atrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Families of Spinal Muscular Atrophy (Other); Leadiant Biosciences, Inc. (Industry); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11893
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2016-08

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy (SMA); Valproic Acid
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Valproic Acid

INTERVENTIONS:
Drug: Valproic Acid

SUMMARY:
This is an open label phase I/II clinical trial to assess safety, tolerability and potential effect on SMN mRNA and protein in vivo of a compound in which preliminary evidence supports a potential effect on SMN levels in vitro.

DETAILED DESCRIPTION:
This is an open label phase I/II trial of valproic acid in 40 SMA subjects > 2 years of age with severe, intermediate, and mild phenotypes. Primary outcome measures includes laboratory and physical examination assessments to monitor effects on liver, hematologic, metabolic and nutritional status. Secondary outcomes includes measures of gross motor function; electrophysiologic measures of denervation; DEXA estimates of body composition, bone mineral density and content; measures of pulmonary function; and quantitative SMN mRNA and protein levels in blood cells. Subjects will need 2-3 baseline visits over a 3 -6 month period prior to enrollment. Follow-up visits will be scheduled at 3, 6 and 12 months on treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of SMA, confirmed by genetic testing
* Only patients 2 years of age and older at enrollment will be eligible

Exclusion Criteria:

* Patients taking any medications with known hepatotoxicity, congenital metabolic disorders or on multiple anticonvulsant medications
* Patients taking medications which may interact with VPA
* Patients on ventilatory support for more than 16 hours per day
* Patients currently enrolled in other treatment trials

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42
Dates: Start 2003-09; Study Completion 2006-02

PRIMARY OUTCOMES:
To assess safety and tolerability of VPA in SMA patients greater than 2 years of age

SECONDARY OUTCOMES:
To look for a potential in vivo effect of VPA on SMN mRNA in patient blood cells at routinely used clinical doses
Measures of gross motor function
Electrophysiologic measures of denervation
DEXA estimates of body composition, bone mineral density and content
Measures of pulmonary function

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn J Swoboda, M.D, Principal Investigator — University of Utah/Primary Children's Medical Center
Locations (1):
- University of Utah/Primary Children's Medical Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Brahe C, Bertini E. Spinal muscular atrophies: recent insights and impact on molecular diagnosis. J Mol Med (Berl). 1996 Oct;74(10):555-62. doi: 10.1007/s001090050059. PMID 8912176
- [Background] Roberts DF, Chavez J, Court SD. The genetic component in child mortality. Arch Dis Child. 1970 Feb;45(239):33-8. doi: 10.1136/adc.45.239.33. PMID 4245389
- [Background] Pearn J. Incidence, prevalence, and gene frequency studies of chronic childhood spinal muscular atrophy. J Med Genet. 1978 Dec;15(6):409-13. doi: 10.1136/jmg.15.6.409. PMID 745211
- [Background] Czeizel A, Hamula J. A hungarian study on Werdnig-Hoffmann disease. J Med Genet. 1989 Dec;26(12):761-3. doi: 10.1136/jmg.26.12.761. PMID 2614795
- [Background] Emery AE. Population frequencies of inherited neuromuscular diseases--a world survey. Neuromuscul Disord. 1991;1(1):19-29. doi: 10.1016/0960-8966(91)90039-u. PMID 1822774
- [Background] Merlini L, Stagni SB, Marri E, Granata C. Epidemiology of neuromuscular disorders in the under-20 population in Bologna Province, Italy. Neuromuscul Disord. 1992;2(3):197-200. doi: 10.1016/0960-8966(92)90006-r. PMID 1483045
- [Background] Pearn J. Classification of spinal muscular atrophies. Lancet. 1980 Apr 26;1(8174):919-22. doi: 10.1016/s0140-6736(80)90847-8. PMID 6103267
- [Background] Bromberg MB, Swoboda KJ. Motor unit number estimation in infants and children with spinal muscular atrophy. Muscle Nerve. 2002 Mar;25(3):445-7. doi: 10.1002/mus.10050. PMID 11870724
- [Background] Swoboda KJ, Prior TW, Scott CB, McNaught TP, Wride MC, Reyna SP, Bromberg MB. Natural history of denervation in SMA: relation to age, SMN2 copy number, and function. Ann Neurol. 2005 May;57(5):704-12. doi: 10.1002/ana.20473. PMID 15852397
- [Background] Crawford TO. From enigmatic to problematic: the new molecular genetics of childhood spinal muscular atrophy. Neurology. 1996 Feb;46(2):335-40. doi: 10.1212/wnl.46.2.335. No abstract available. PMID 8614490
- [Background] Gilliam TC, Brzustowicz LM, Castilla LH, Lehner T, Penchaszadeh GK, Daniels RJ, Byth BC, Knowles J, Hislop JE, Shapira Y, et al. Genetic homogeneity between acute and chronic forms of spinal muscular atrophy. Nature. 1990 Jun 28;345(6278):823-5. doi: 10.1038/345823a0. PMID 1972783
- [Background] Melki J, Lefebvre S, Burglen L, Burlet P, Clermont O, Millasseau P, Reboullet S, Benichou B, Zeviani M, Le Paslier D, et al. De novo and inherited deletions of the 5q13 region in spinal muscular atrophies. Science. 1994 Jun 3;264(5164):1474-7. doi: 10.1126/science.7910982.
- [Background] Monani UR, Lorson CL, Parsons DW, Prior TW, Androphy EJ, Burghes AH, McPherson JD. A single nucleotide difference that alters splicing patterns distinguishes the SMA gene SMN1 from the copy gene SMN2. Hum Mol Genet. 1999 Jul;8(7):1177-83. doi: 10.1093/hmg/8.7.1177. PMID 10369862
- [Background] Campbell L, Potter A, Ignatius J, Dubowitz V, Davies K. Genomic variation and gene conversion in spinal muscular atrophy: implications for disease process and clinical phenotype. Am J Hum Genet. 1997 Jul;61(1):40-50. doi: 10.1086/513886. PMID 9245983
- [Background] Lefebvre S, Burlet P, Liu Q, Bertrandy S, Clermont O, Munnich A, Dreyfuss G, Melki J. Correlation between severity and SMN protein level in spinal muscular atrophy. Nat Genet. 1997 Jul;16(3):265-9. doi: 10.1038/ng0797-265. PMID 9207792
- [Background] Monani UR, Sendtner M, Coovert DD, Parsons DW, Andreassi C, Le TT, Jablonka S, Schrank B, Rossoll W, Prior TW, Morris GE, Burghes AH. The human centromeric survival motor neuron gene (SMN2) rescues embryonic lethality in Smn(-/-) mice and results in a mouse with spinal muscular atrophy. Hum Mol Genet. 2000 Feb 12;9(3):333-9. doi: 10.1093/hmg/9.3.333. PMID 10655541
- [Background] Feldkotter M, Schwarzer V, Wirth R, Wienker TF, Wirth B. Quantitative analyses of SMN1 and SMN2 based on real-time lightCycler PCR: fast and highly reliable carrier testing and prediction of severity of spinal muscular atrophy. Am J Hum Genet. 2002 Feb;70(2):358-68. doi: 10.1086/338627. Epub 2001 Dec 21. PMID 11791208
- [Background] Mailman MD, Heinz JW, Papp AC, Snyder PJ, Sedra MS, Wirth B, Burghes AH, Prior TW. Molecular analysis of spinal muscular atrophy and modification of the phenotype by SMN2. Genet Med. 2002 Jan-Feb;4(1):20-6. doi: 10.1097/00125817-200201000-00004. PMID 11839954
- [Background] Fischer U, Liu Q, Dreyfuss G. The SMN-SIP1 complex has an essential role in spliceosomal snRNP biogenesis. Cell. 1997 Sep 19;90(6):1023-9. doi: 10.1016/s0092-8674(00)80368-2. PMID 9323130
- [Background] Chang JG, Hsieh-Li HM, Jong YJ, Wang NM, Tsai CH, Li H. Treatment of spinal muscular atrophy by sodium butyrate. Proc Natl Acad Sci U S A. 2001 Aug 14;98(17):9808-13. doi: 10.1073/pnas.171105098. PMID 11504946
- [Background] Andreassi C, Jarecki J, Zhou J, Coovert DD, Monani UR, Chen X, Whitney M, Pollok B, Zhang M, Androphy E, Burghes AH. Aclarubicin treatment restores SMN levels to cells derived from type I spinal muscular atrophy patients. Hum Mol Genet. 2001 Nov 15;10(24):2841-9. doi: 10.1093/hmg/10.24.2841. PMID 11734549
- [Background] Brichta L, Hofmann Y, Hahnen E, Siebzehnrubl FA, Raschke H, Blumcke I, Eyupoglu IY, Wirth B. Valproic acid increases the SMN2 protein level: a well-known drug as a potential therapy for spinal muscular atrophy. Hum Mol Genet. 2003 Oct 1;12(19):2481-9. doi: 10.1093/hmg/ddg256. Epub 2003 Jul 29. PMID 12915451
- [Background] Andreassi C, Angelozzi C, Tiziano FD, Vitali T, De Vincenzi E, Boninsegna A, Villanova M, Bertini E, Pini A, Neri G, Brahe C. Phenylbutyrate increases SMN expression in vitro: relevance for treatment of spinal muscular atrophy. Eur J Hum Genet. 2004 Jan;12(1):59-65. doi: 10.1038/sj.ejhg.5201102. PMID 14560316
- [Background] Bohmer T, Rydning A, Solberg HE. Carnitine levels in human serum in health and disease. Clin Chim Acta. 1974 Nov 20;57(1):55-61. doi: 10.1016/0009-8981(74)90177-6. No abstract available. PMID 4279150
- [Background] Brooks H, Goldberg L, Holland R, Klein M, Sanzari N, DeFelice S. Carnitine-induced effects on cardiac and peripheral hemodynamics. J Clin Pharmacol. 1977 Oct;17(10 Pt 1):561-8. doi: 10.1177/009127007701701003. No abstract available. PMID 915022
- [Background] Christiansen RZ, Bremer J. Active transport of butyrobetaine and carnitine into isolated liver cells. Biochim Biophys Acta. 1976 Nov 2;448(4):562-77. doi: 10.1016/0005-2736(76)90110-3. PMID 974147
- [Background] Lindstedt S, Lindstedt G. Distribution and Excretion of Carnitine in the Rat. Acta. Chem. Scand. 1961; 15:701-702
- [Background] Rebouche CJ, Engel AG. Carnitine metabolism and deficiency syndromes. Mayo Clin Proc. 1983 Aug;58(8):533-40. PMID 6348429
- [Background] Rebouche CJ, Paulson DJ. Carnitine metabolism and function in humans. Annu Rev Nutr. 1986;6:41-66. doi: 10.1146/annurev.nu.06.070186.000353. PMID 3524622
- [Background] Igarashi N, Sato T, Kyouya S. Secondary carnitine deficiency in handicapped patients receiving valproic acid and/or elemental diet. Acta Paediatr Jpn. 1990 Apr;32(2):139-45. doi: 10.1111/j.1442-200x.1990.tb00799.x. PMID 2143048
- [Background] Thurston JH, Hauhart RE. Amelioration of adverse effects of valproic acid on ketogenesis and liver coenzyme A metabolism by cotreatment with pantothenate and carnitine in developing mice: possible clinical significance. Pediatr Res. 1992 Apr;31(4 Pt 1):419-23. doi: 10.1203/00006450-199204000-00023. PMID 1570210
- [Background] Tein I, DiMauro S, Xie ZW, De Vivo DC. Valproic acid impairs carnitine uptake in cultured human skin fibroblasts. An in vitro model for the pathogenesis of valproic acid-associated carnitine deficiency. Pediatr Res. 1993 Sep;34(3):281-7. doi: 10.1203/00006450-199309000-00008. PMID 8134167
- [Background] Melegh B, Pap M, Morava E, Molnar D, Dani M, Kurucz J. Carnitine-dependent changes of metabolic fuel consumption during long-term treatment with valproic acid. J Pediatr. 1994 Aug;125(2):317-21. doi: 10.1016/s0022-3476(94)70218-7. PMID 8040784
- [Background] Tein I, Xie ZW. Reversal of valproic acid-associated impairment of carnitine uptake in cultured human skin fibroblasts. Biochem Biophys Res Commun. 1994 Oct 28;204(2):753-8. doi: 10.1006/bbrc.1994.2523. PMID 7980539
- [Background] Van Wouwe JP. Carnitine deficiency during valproic acid treatment. Int J Vitam Nutr Res. 1995;65(3):211-4. PMID 8830002
- [Background] Evangeliou A, Vlassopoulos D. Carnitine metabolism and deficit--when supplementation is necessary? Curr Pharm Biotechnol. 2003 Jun;4(3):211-9. doi: 10.2174/1389201033489829. PMID 12769764
- [Background] Coulter DL. Carnitine deficiency: a possible mechanism for valproate hepatotoxicity. Lancet. 1984 Mar 24;1(8378):689. doi: 10.1016/s0140-6736(84)92209-8. No abstract available. PMID 6142383
- [Background] Coulter DL. Carnitine, valproate, and toxicity. J Child Neurol. 1991 Jan;6(1):7-14. doi: 10.1177/088307389100600102. PMID 2002205
- [Background] Scriver C, Beautet A, Sly W ,Valle D. The Metabolic Basis of Inherited Disease. New York: McGraw Hill,1989
- [Background] Schaub J, Van Hoof F, Vis H.Inborn Errors of Metabolism. New York:Raven Press, 1991
- [Background] Standardization of Spirometry, 1994 Update. American Thoracic Society. Am J Respir Crit Care Med. 1995 Sep;152(3):1107-36. doi: 10.1164/ajrccm.152.3.7663792. No abstract available.
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Derived] Swoboda KJ, Scott CB, Reyna SP, Prior TW, LaSalle B, Sorenson SL, Wood J, Acsadi G, Crawford TO, Kissel JT, Krosschell KJ, D'Anjou G, Bromberg MB, Schroth MK, Chan GM, Elsheikh B, Simard LR. Phase II open label study of valproic acid in spinal muscular atrophy. PLoS One. 2009;4(5):e5268. doi: 10.1371/journal.pone.0005268. Epub 2009 May 14. PMID 19440247